CLINICAL TRIAL: NCT01793779
Title: Comparison of Pre-exercise Beta-hydroxy-beta-methylbutyrate Free Acid (HMB-FA) and Cold Water Therapy for the Attenuation of Muscle Damage and Soreness in Experienced Resistance Trained Individuals.
Brief Title: Comparison of Pre-exercise Beta-hydroxy-beta-methylbutyrate Free Acid (HMB-FA) and Cold Water Therapy for the Attenuation of Muscle Damage and Soreness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Metabolic Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: MTI2013-CS01
Record Dates: First submitted 2013-02-13; First posted 2013-02-18 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: Muscle Damage

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Placebo Comparator): Placebo supplement given prior to exercise and two times per day following exercise
  Interventions: Dietary Supplement: Placebo
- cold water immersion (Experimental): Placebo supplement to be give prior to exercise and two times per day following exercise in combination with cold water immersion therapy following exercise
  Interventions: Procedure: cold water immersion; Dietary Supplement: Placebo
- HMB-FA (Experimental): beta-hydroxy-beta-methylbutyrate free acid supplement to be give prior to exercise and two times per day following exercise
  Interventions: Dietary Supplement: beta-hydroxy-beta-methylbutyrate free acid (HMB-FA)
- cold water immersion group + HMB-FA (Experimental): beta-hydroxy-beta-methylbutyrate free acid supplement give prior to exercise and two times per day following exercise in combination with cold water immersion therapy following exercise
  Interventions: Procedure: cold water immersion; Dietary Supplement: beta-hydroxy-beta-methylbutyrate free acid (HMB-FA)

INTERVENTIONS:
Procedure: cold water immersion
  Arms: cold water immersion; cold water immersion group + HMB-FA
Dietary Supplement: beta-hydroxy-beta-methylbutyrate free acid (HMB-FA)
  Arms: HMB-FA; cold water immersion group + HMB-FA
Dietary Supplement: Placebo
  Arms: Control; cold water immersion

SUMMARY:
Study Objectives

1. Compare beta-hydroxy-beta-methylbutyrate free acid (HMB-FA) to cold water immersion on performance recovery from an acute bout of high intensity resistance exercise.
2. Compare HMB-FA + Cold water immersion to HMB-FA or cold water immersion.
3. Examine the effect of these recovery modalities on markers of muscle damage, inflammation and immune function.

Subjects

Subjects (men and women, 18 - 35 y) with at least one year of resistance training experience will be recruited. Subjects will be randomly divided into one of four groups: a cold water immersion group (CW), HMB-FA, CW+HMB-FA and a control group (CT).

Study Protocol

Subjects will report to the Human Performance Laboratory (HPL) on four separate occasions. On the first visit (T1) subjects will be tested for maximal strength [one repetition-maximum (1-RM)] on the squat, dead lift and barbell lunge exercises.] On their second visit (T2) subjects will perform a lower body resistance exercise session consisting of four sets of the squat, dead lift and barbell lunge exercises. All subjects will then report back to the HPL at 24- (T3) and 48-hours (T4) post-exercise. During T3 and T4, subjects will perform four sets of the squat exercise only using the same loading pattern and rest interval length as T2. Following the T2 and T3 workouts subjects in CT will undergo no treatment; subjects in CW will be required to sit in a whirlpool tub for 10-min up to their umbilicus in water at 50° F - 54° F (10° C - 12° C); subjects in HMB-FA will be provided the supplement 30 min prior each workout and CW+HMB-FA will be administered together at time points describe above.

Statistical Analysis

Statistical evaluation of performance and biochemical changes will be accomplished using a repeated measures analysis of variance (ANOVA).

ELIGIBILITY:
Inclusion Criteria:

* At least one-year of resistance training experience
* Free of any physical limitations (determined by health and activity questionnaire).
* Between the ages of 18 and 35

Exclusion Criteria:

* Inability to perform physical exercise (determined by health and activity questionnaire)
* Taking any other nutritional supplement or performance enhancing drug (determined from health and activity questionnaire).
* Any chronic illness that causes continuous medical care
* Taking any type of prescription or over-the-counter medication, having any chronic illness causing you to seek medical care, pregnancy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Maximal muscle strength | Change from baseline over 48 hours post-exercise.
  The 1-RM tests will be performed to assess maximal muscle strength.

SECONDARY OUTCOMES:
Muscle damage | Change from baseline over 48 hours post-exercise.
  Serum creatine kinase and myoglobin concentrations will be analyzed as markers of muscle damage.

OTHER OUTCOMES:
Muscle soreness | Change from baseline over 48-hours post-exercise.
  Subjects will be asked to rate their degree of lower body muscle soreness using a 15-cm visual analog scale (VAS).
Lower body power | Change from baseline over 48 hours post-exercise.
  Lower body power during the squat exercise protocol will be measured each repetition with a Tendo™ Power Output Unit.
Immune Markers | Change from baseline over 48 hours post-exercise.
  Immune (IL-6, IL-10, Macrophage inflammatory protein-1β, tumor necrosis factor-α) markers will be analyzed.
C-reactive protein | Change from baseline over 48 hours post-exercise.
  The Inflammatory marker, C-reactive protein, will be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Florida, Sport and Exercise Science, Orlando, Florida, United States

REFERENCES:
- [Background] Ascensao A, Leite M, Rebelo AN, Magalhaes S, Magalhaes J. Effects of cold water immersion on the recovery of physical performance and muscle damage following a one-off soccer match. J Sports Sci. 2011 Feb;29(3):217-25. doi: 10.1080/02640414.2010.526132. PMID 21170794
- [Background] Fuller JC Jr, Sharp RL, Angus HF, Baier SM, Rathmacher JA. Free acid gel form of beta-hydroxy-beta-methylbutyrate (HMB) improves HMB clearance from plasma in human subjects compared with the calcium HMB salt. Br J Nutr. 2011 Feb;105(3):367-72. doi: 10.1017/S0007114510003582. Epub 2010 Dec 7. PMID 21134325